CLINICAL TRIAL: NCT03867825
Title: Hemodynamic Monitoring of Newborn Infants With Impedance Cardiography Versus Echocardiography; a Validation Study
Status: Withdrawn | Type: Observational
Why Stopped: Never got medical equipment that worked properly
Sponsor: University Hospital of North Norway (Other)
Collaborators: Knut Helge Kaspersen, MD (Unknown); Per Ivar Kaaresen, MD, PhD (Unknown); Nils Thomas Songstad, MD, PhD (Unknown); Ganesh Acharya, Professor (Unknown)
Responsible Party: Principal Investigator, Claus Klingenberg, Professor, University Hospital of North Norway
Other Study IDs: 2014/2312
Record Dates: First submitted 2019-03-06; First posted 2019-03-08 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Hemodynamics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Non-invasive hemodynamic monitoring — Impedance cardiography

SUMMARY:
Background:

Impedance cardiography (ICG) is a noninvasive method for continuous left cardiac output monitoring based on measurement of thoracic electrical bioimpedance. The objective of this study is to validate an ICG device by investigating the agreement in cardiac output (CO; left ventricular output x heart rate) measurements performed by ICG and echocardiography. The ICG device (PhysioFlow) has a new filter technology reducing signal noise and enabling measurements in patients who are moving freely.

Material and Methods

* Design: Prospective observational study.
* Inclusion: 30 healthy term infants between 24 and 48 hours of age, after parental consent
* Methods: Continuous measurement with ICG over a 30 min period and point of care echocardiography
* Primary outcome: Agreement (bis and precision) between measurement of CO with ICG and echocardiography.
* Secondary outcomes: Agreement between other echocardiographic indices of myocardial function and ICG parameters (early diastolic filling ratio, cardiac index, ventricular ejection time and left cardiac work index).
* Statistics: Agreement between ICG and echocardiography data will be evaluated using Bland-Altman statistics, including the calculation of mean bias (average difference between measurements) with corresponding standard deviation and lower and upper limits of agreements (95% confidence interval).

ELIGIBILITY:
Inclusion Criteria:

* Newborn infants

Exclusion Criteria:

* Infants > 1 month of age

Max Age: 1 Month | Sex: All
Age Groups: Child
Study Population: Term healthy infants
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Cardiac output | one hour
  Stroke volume x heart rate